CLINICAL TRIAL: NCT02815774
Title: A Parallel, Open Phase Ih Study to Access the Pharmacokinetic of SP2086 in Renal Insufficiency Patients
Brief Title: SP2086 Pharmacokinetic Study in Renal Insufficiency Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-SP2086-Ih
Record Dates: First submitted 2016-01-03; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Renal Insufficiency
Keywords: SP2086; Renal Insufficiency; Pharmacokinetic
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- health volunteers (Active Comparator): this group patients were given SP2086 50mg only one time.
  Interventions: Drug: SP2086
- mild renal insufficiency (Active Comparator): this group patients were given SP2086 50mg only one time.
  Interventions: Drug: SP2086
- moderate renal insufficiency (Active Comparator): this group patients were given SP2086 50mg only one time.
  Interventions: Drug: SP2086
- severe renal insufficiency (Active Comparator): this group patients were given SP2086 50mg only one time.
  Interventions: Drug: SP2086
- end-stage renal insufficiency (Active Comparator): this group patients were given SP2086 50mg only one time.
  Interventions: Drug: SP2086

INTERVENTIONS:
Drug: SP2086 — all subjects were given SP2086 50mg only one time.

SUMMARY:
The purpose of the study is to investigate the SP2086 pharmacokinetic in Renal Insufficiency Patients.

DETAILED DESCRIPTION:
This trial adopt in a parallel, open, single dose study design. The subject was divided into one of five groups according to the degree of renal Insufficiency, which including normal, mild, moderate, severe, and end-stage. All subjects were given SP2086 50mg, and collected the blood samples before and after the medicine taken.

ELIGIBILITY:
Inclusion Criteria:

* with a body mass index(BMI) between 19 and 28 Kg/m2;Weight:≥50Kg(male),≥45kg(female)
* The endogenous creatinine clearance of subjects in groups must meet the standards of Ccr in renal function in installment:mild renal insufficiency:60-89 - ml/min;Moderate renal insufficiency: 30 to 59 ml/min;Severe renal insufficiency: 15-29 ml/min;End-stage renal disease: < 15 ml/min.Normal renal function: 90 ml/min or more.
* Had signed the informed consent himself or herself voluntarily.

Exclusion Criteria:

* Cannot tolerate oral medicine.
* Not control or unstable cardiovascular, respiratory, liver, digestive, endocrine, hematopoietic, the mental or nerve system diseases.
* Had the digestive surgery that could affect drug absorption.
* The clinical significance of arrhythmia.
* Acute hepatitis, chronic liver disease; ALT or AST value was 2 times greater than upper normal limit, Total bilirubin value was 1.5 times greater than upper normal limit.
* HBV surface antigen, HCV antibody, or HIV antibody was positive.
* history of drug allergy or allergic constitution or family history of allergy.
* Had Used hormonal contraception within 3 months;
* Had Used DPP - IV inhibitor within 2 weeks;
* Had Used traditional Chinese medicine (Chinese herbs, Chinese patent medicine) within 2 weeks;
* Had Used acid inhibitors within 2 weeks;
* Alcohol, tobacco, drug abusers;alcohol abuse is defined as a day for regular alcohol consumption more than the following standards: beer 570 ml, light beer 750 ml, red wine 200 ml, white wine 60 ml, which including about 20g alcohol;Tobacco is defined as five or more per day.
* 2 days before the randomization till to the end ,the patients can not ban alcohol, tobacco, or reference food or drink containing caffeine or xanthine , or vigorous exercise, or there are other factors that can affect drug absorption, distribution, metabolism and excretion
* The patient had participated three times or more clinical trial in one year, or one time within 3 months.
* Pregnancy or lactation women, or a fertility male or female is not willing to contraception during test.
* History of blood donation or participate in blood donation, or by blood transfusion in 3 months prior to screening.
* Researchers considered that there was any situation that may cause the participants can't finish this study or bring any obvious risk to subjects.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to 96 hours
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086
The maximum plasma concentration (Cmax) of SP2086 acid | up to 96 hours
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086
The area under the plasma concentration-time curve (AUC) of SP2086 | up to 96 hours
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086
The area under the plasma concentration-time curve (AUC) of SP2086 acid | up to 96 hours
  AUC (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jia Miao, P.H.D, Principal Investigator — West China Hospital